CLINICAL TRIAL: NCT03657693
Title: MRI for Quantitative Measurement of Pulmonary Growth and Development in Term and Extremely Pre-Term Babies in the BPD Center of Excellence
Brief Title: MRI in BPD Subjects
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_BPD_COE_001
Record Dates: First submitted 2018-05-16; First posted 2018-09-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and remnant blood and BAL samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- BPD: Infants born premature requiring oxygen
  Interventions: Diagnostic Test: NICU MRI; Diagnostic Test: Polysomnography
- Controls
  Interventions: Diagnostic Test: NICU MRI; Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: NICU MRI — MRI device that is not FDA approved.
Diagnostic Test: Polysomnography — Polysomnography to better determine obstruction index in the airway.

SUMMARY:
The investigators are wanting to learn more about early development of the lungs and to help them better understand prematurity and the development of a breathing disorder call BPD (Bronchopulmonary Dysplasia)

DETAILED DESCRIPTION:
This is an observational case study involving up to three MRI visits. The first MRI will be complete after the infant's clinical initial evaluation. The second image will be obtained approximately 1 month later and the third MRI will be complete prior to discharge. Infants will be imaged at various ages, based up their initial evaluation. The investigators will collect urine and obtain clinically collected remnant blood around time of MRI, tracheal/endotracheal aspirate at time of the MRI when available and BAL samples as clinically available. MRI findings will be correlated with laboratory findings and outcomes from the medical record, and a research database will be built for the data. The investigators will also obtain a one-time MRI visit in non-BPD NICU patients to acquire data related to normal vasculature and pulmonary alveolar development.

Sub-study 1: Inpatient polysomnography Patients with the same inclusion/exclusion criteria as reported below will be approached for a brief inpatient polysomnogram. The population will include patients with and without BPD. The polysomnography (PSG) will be performed in the NICU within 1 week from the MRI that is obtained prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* any term age NICU patient

Exclusion Criteria:

* - ECMO,
* Evidence of congenital diseases that may affect lung development, such as congenital diaphragmatic hernia,
* Suspected muscular dystrophy or neurologic disorder that may affect lung development.
* Significant genetic or chromosomal abnormalities that may affect lung development
* Evidence of any respiratory infection at the time of imaging (imaging may be rescheduled for a common viral infection such as a cold).
* Standard MRI exclusion criteria as set forth by the CCHMC Department of Radiology. This includes any contraindications from tracheostomy tubes that are not MR compatible.

Max Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Bronchopulmonary Dysplasia (BPD)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Anatomic phenotypes using MRI | baseline
  Investigate parenchymal and vascular structures, regional cardiopulmonary function, and dynamic airway collapse in BPD infants during quiet unsedated breathing.

SECONDARY OUTCOMES:
Polysomnography | within a week of baseline MRI
  Determine the correlation between upper airway MRI and the obstruction index in the polysomnography.

OTHER OUTCOMES:
Change in the anatomic phenotype using MRI | 1 month post baseline and discharge from NICU
  Compare the parenchymal reader scoring, cardiac analysis, and airway scoring over the span of the BPD infant's time in the NICU.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Megan Schmitt, Cincinnati, Ohio, United States